CLINICAL TRIAL: NCT04325529
Title: Novel Treatment Targets For Affective Disorders Through Cross-Species Investigation of Approach/Avoidance Decision Making
Brief Title: Pharmaco-Neuroimaging Studies of Approach/Avoidance Behaviors and Post-Mortem Studies: Study 1.2 (Stress Manipulation)
Status: Active, not recruiting | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Diego Pizzagalli, Principal Investigator; Professor, Department of Psychiatry, Harvard Medical School, Mclean Hospital, Mclean Hospital
Other Study IDs: 2020A000886
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Major Depression in Remission

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- remitted MDD: Unmedicated Remitted Participants with Past History of MDD
  Interventions: Device: Aversive stimuli
- Control subjects: healthy control subjects
  Interventions: Device: Aversive stimuli

INTERVENTIONS:
Device: Aversive stimuli — Electrotactile stimulation will be used as the aversive stimulus. The aversive stimulus is delivered in the form of a mild half-second stimulation to the ankle, calibrated to a subjective threshold that is uncomfortable but not painful. This stimulation is delivered by Digitimer DS8R Constant Current Stimulator (Digitimer North America, LLC. Ft. Lauderdale, FL). Its previous model DS71 has been safely implemented in studies with previously MGH-approved IRB's (Milad et al., 2013).
  Other Names: no other name

SUMMARY:
This study investigates how remitted individuals with past major depressive disorder (MDD) make approach-avoidance decisions and which brain regions are implicated in such decisions. Information collected through MRI and behavioral tasks will be used to predict depressive symptoms in the future.

DETAILED DESCRIPTION:
The overarching goals of this research are to investigate: (1) neural substrates of approach/avoidance behaviors in remitted MDDs; (2) stress-induced signaling in remitted individuals with past MDD; (3) neural markers that prospectively predict disease course.

This will be achieved through an innovative method of using functional magnetic resonance imaging (fMRI) during an approach/avoidance decision-making task.

ELIGIBILITY:
Inclusion Criteria for all participants:

* All genders, races, and ethnic origins, aged between 18 and 45
* Capable of providing written informed consent, and fluent in English
* Right-handed
* Absence of any psychotropic medications for at least 2 weeks
* Has a smartphone (iPhone or Android) (needed for Ecological Momentary Assessment)

Inclusion Criteria for "Remitted MDD" group:

* Meets inclusion criteria for all subjects, plus:
* History of MDD as defined by DSM-5
* Absence of anxiety disorder for the past two months

Exclusion Criteria for all participants:

* Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment
* Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, IUD, s/p tubal ligation, or partner with vasectomy)
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder
* History of psychiatric illnesses, other than depression or anxiety disorders among the Current MDD and Remitted MDD groups
* History of substance use disorder or alcohol use disorder (as these terms are defined by DSM-5); except depressed subjects may have a history of 'Mild' substance/alcohol use disorder only if it ended as least 12 months ago
* History of cocaine or stimulant use or dopaminergic drugs
* History or current diagnosis of dementia, or a score of < 26 on the Mini Mental State Examination at the screening visit;
* Patients with mood congruent or mood incongruent psychotic features
* Current use of other psychotropic drugs
* Clinical or laboratory evidence of hypothyroidism
* Patients with a lifetime history of electroconvulsive therapy (ECT)
* Failure to meet standard MRI safety requirements
* Abnormal ECG and lab results
* History of seizure disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The subjects for this research will be 96 participants recruited from the community by the Center for Depression, Anxiety and Stress Research (Director: Dr. Diego Pizzagalli, Ph.D.). Participants will include: (1) 48 participants with past MDD; and (2) 48 demographically matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Interview | Baseline
  For assessing psychological state
Behavioral Performance on the Probabilistic Reward Task (PRT) | Baseline
  The Probablilistic Reward Task assesses positive reinforcement learning.
MRI Data | MRI scans take place within 30 days of Screening Visit
  For testing the neural correlates of approach-avoidance decision making behaviors in a trans-diagnostic sample
Salivary Cortisol | Baseline
  For assessing stress level
Follow-up Clinical interviews | Change from Baseline at 6 months and 12 months after the MRI scanning visit
  To assess psychological state changes

CONTACTS AND LOCATIONS:
Overall Officials: Diego Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided